CLINICAL TRIAL: NCT00467272
Title: Phase II, Open-Label Study to Evaluate the Safety and Efficacy of Daptomycin in the Treatment of Catheter-Related Gram Positive Bloodstream Infections
Brief Title: Catheter Related - Gram Positive Bloodstream Infections
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Cubist Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0958
Record Dates: First submitted 2007-04-26; First posted 2007-04-30 (Estimated); Results first posted 2021-02-08 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-01

CONDITIONS: Bloodstream Infection
Keywords: Catheter-Related Bloodstream Infections; Bloodstream Infection; Daptomycin; Cubicin; CRBSI
MeSH Terms: conditions — Sepsis | interventions — Daptomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Daptomycin (Experimental): Daptomycin 6 mg/kg intravenous (IV) every 24 hours for at least 7-14 days, depending on the type of bacteria.
  Interventions: Drug: Daptomycin

INTERVENTIONS:
Drug: Daptomycin — 6 mg/kg IV every 24 hours for at least 7-14 days, depending on the type of bacteria. Treatment expected to be at least 14 days for SA and at least 7 days for enterococci and CNS, Corynebacterium, and Propionibacterium.
  Other Names: Cubicin

SUMMARY:
Primary Objective:

-Evaluate the clinical efficacy and safety of Daptomycin given for treatment of catheter-related bloodstream infections (CRBSI) due to gram positive bacteremia in the context of standard of care antimicrobial therapy consisting mainly of Vancomycin with or without initial treatment with beta lactam antibiotics.

DETAILED DESCRIPTION:
THE STUDY DRUG:

Daptomycin is an antibiotic designed to treat a variety of bacterial infections that are difficult to treat.

STUDY TREATMENT:

If you are found to be eligible to take part in this study, you will be given daptomycin by vein over 30 minutes every 24 hours for at least 7-14 days, depending on the type of bacteria that you have.

The central venous catheter (CVC) will either be removed, or it will be exchanged over a guide wire. The decision to remove or exchange the CVC and timing of the placement of the CVC will be decided by your primary physician and the willingness of you to remove or exchange your infected CVC. This will be done within 96 hours after your first positive blood culture (first blood drawn that showed bacteria). A CVC is a sterile flexible tube that will be placed into a large vein while you are under local anesthesia. Your doctor will explain this procedure to you in more detail, and you will be required to sign a separate consent form for this procedure.

If the study doctor and/or your primary doctor suspects that you have a mixed infection (2 or more certain types of bacteria) or pneumonia, you will also be treated with different types of antibiotics, by vein or mouth, in combination with the study drug. These antibiotics may include aztreonam, cefepime, imipenem, meropenem, ciprofloxacin hydrochloride, bactrim, and/or amoxicillin/clavulanate (a combination antibiotic).

If you are discharged from the hospital before completing the study medication, arrangements will be made to provide infusions on an outpatient basis (by a nurse, yourself, or a family member). You and/or a family member will be taught (by a nurse) how to take the study medication at home. Before you are discharged from the hospital, you will receive the kits that include enough supplies for you and/or a family member to give daptomycin by vein. If medication will be given at home, a prescription will be given to you to pick up your medication from the pharmacy before you discharge from the hospital. If possible, your primary doctor may arrange for you to receive medication at the M. D. Anderson outpatient treatment center, or a nurse will be scheduled to visit you at home to give you the medication.

STUDY TESTS/PROCEDURES:

During each week of treatment, you will have the following exams/procedures performed once a week.

* You will have blood drawn (about 1 tablespoon) for routine tests. It may be drawn from the CVC, if the CVC is still in place. The CVC exit site will be examined at each visit until you have no more signs or symptoms of infection.
* You will also have blood drawn (about 1 tablespoon) for a blood culture every other day until it no longer shows signs of infection.
* You will be asked about any symptoms or illnesses that you may have experienced since your last visit.

LENGTH OF STUDY:

Participation on this study will last for no more than 60 days (about 2 months).

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating females with an age of greater than or equal to 18 years.
* The suspected culprit on exchangeable central venous catheter (CVC) is tunneled or non-tunnel (including ports and PICC) and antibiotic or non-antibiotic coated catheter inserted in the subclavian, jugular, peripheral or femoral vein.
* Patients must have at least two signs of sepsis from the list below, in any combination, within 48 hours prior to Daptomycin therapy and no other source for the bacteremia other than CVC: a. Core temperature =/>38.0 degrees C or =/<36.0 degrees C, measured orally, rectally, tympanic ally or via a central catheter. If auxiliary add 0.5 degrees C to the measured temperature; b. Pulse rate =/> 100 beats/min.; c. Respiratory rate =/> 20/min.; d. white blood cell (WBC) count =/>12,000/mm^3 or =/<4,000/mm^3 differential count showing >10% band forms; e. Systolic blood pressure =/<90 mm Hg.
* Patients with probable or definite diagnosis of uncomplicated CVC-related gram positive bacteremia that includes at least one positive blood culture for Coagulase Negative Staphylococci (CNS), Staphylococcus aureus (SA), Enterococci, Corynebacterium, and Propionibacterium (If the positive blood culture is drawn through the CVC for skin flora such as CNS, Corynebacterium, Propionibacterium, Micrococcus and Bacillus, then at least >15 colonies/ml will be required or the time of positive (DTP) of CVC at least 2 hours earlier than the peripheral culture).
* Signed informed consent.
* No apparent source for the clinical manifestation of bacteremia other than the catheter (may have local signs and symptoms at the catheter site).

Exclusion Criteria:

* Estimated Serum Creatinine Clearance <30 mL/min (according to Cock-Gault-formula)at the time gram positive bacteremia was diagnosed unless the patient is on dialysis.
* Bilirubin >4 times the upper limit of normal at the time gram positive bacteremia was diagnosed.
* Treatment with an antibiotic, such as vancomycin, linezolid, tigecycline or daptomycin, effective against resistant gram positive bacterial infections, such as methicillin resistant staphylococci, for more than 48 hours within 72 hours of study medication initiation, unless treatment failed that is defined as a persistent fever, leukocytosis, and/or repeated positive blood cultures (CVC and peripheral) for 72 hours or longer of appropriate antibiotics treatment other than Daptomycin.
* Documented gram positive bacteremia within last 1 month due to source other than CVC.
* Patients who have participated in another investigational anti-infective study within 30 days.
* History of hypersensitivity to lipopeptides.
* Presence of additional source of infection with same organism cultured from blood, eg. endocarditis (as evidenced by vegetations on an echocardiogram), septic thrombosis.
* Conditions with markedly decreased albumin in plasma (<1.5 g/dl), e.g., cirrhosis, nephritic syndrome, end-stage renal disease.
* Prosthetic valve.
* Oliguria defined as urine output of <20 cc/hour averaged over 24 hours.
* Possible complicated CRBSI with persistent bacteremia for more than 48 hours on active antimicrobial therapy (such as osteomyelitis, endocarditis, and septic thrombosis).
* Patients with diagnosis of pneumonia that is due to S. aureus organism, e.g, S. aureus from sputum or bronchial cultures.
* creatine phosphokinase (CPK) >10 times max-normal in asymptomatic patients and CPK >5 max-normal in symptomatic patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-03; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Issam Raad, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: June 2006 to March 2008. All recruitment done at UT MD Anderson Cancer Center.
Pre-assignment Details: This study is the continuation of trial NCT00507247 which included 11 participants; the results has been combined NCT00507247 and NCT00467272. A total of combined participants were 41, out of which 38 participants were included in the analysis and 3 participants were excluded.
Groups:
- Daptomycin 6 mg/kg IV: Daptomycin: 6 mg/kg IV every 24 hours for at least 7-14 days, depending on the type of bacteria. Treatment expected to be at least 14 days for Staphylococcus aureus (SA) and at least 7 days for enterococci and Coagulase Negative Staphylococci (CNS), Corynebacterium and Propionibacterium.
Period: Overall Study
Arm/Group | Daptomycin 6 mg/kg IV
Started | 41
Completed | 38
Not Completed | 3
Not completed — Pneumonia | 2
Not completed — Thrombophlebitis | 1

BASELINE CHARACTERISTICS:
Population: 40 participants were enrolled in the daptomycin arm. The analysis included 38 participants who received Daptomycin: 3 participants were excluded from analysis prior to study entry.
Arm/Group | Daptomycin 6 mg/kg IV
Number analyzed (Participants) | 38
Age, Continuous [Median (Full Range); unit: years] | 53 [17 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 25
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response Within 48 Hours
Description: Number of participants with clinical response within 48 hours from initiation of Daptomycin, estimated by Bayesian posterior credible interval. Clinical response defined as resolution of clinical signs and symptoms within 48 hours from initiating the study drug.
Time Frame: Within 48 hours from initiating the study drug
Population: Of the 38 participants analyzed, one participant was excluded from the analyses because the date of symptom resolution was missing.
Measure: Count of Participants; unit: Participants
Arm/Group | Daptomycin 6 mg/kg IV
Number analyzed (Participants) | 37
Participants | 28

2. Primary Outcome: Clinical Response Within 7 Days
Description: Number of participants with clinical response within 1 week from initiation of Daptomycin, estimated by Bayesian posterior credible interval. Clinical response defined as resolution of clinical signs and symptoms within 7 days from initiating the study drug.
Time Frame: Within 7 days from initiating the study drug
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Daptomycin 6 mg/kg IV
Number analyzed (Participants) | 37
Participants | 33

3. Primary Outcome: Microbiological Response Within 48 Hours
Description: Number of participants with microbiological response within 48 hours from initiation of Daptomycin. Microbiological response defined as eradication of the microorganism from the bloodstream (negative blood cultures).
Time Frame: Within 48 hours from initiating the study drug
Population: Of the 38 participants analyzed, one participant was excluded from the analyses because the date of microbiological eradication was unknown.
Measure: Count of Participants; unit: Participants
Arm/Group | Daptomycin 6 mg/kg IV
Number analyzed (Participants) | 37
Participants | 29

4. Primary Outcome: Microbiological Response Within 7 Days
Description: Number of participants with microbiological response within 7 days from initiation of Daptomycin. Microbiological response defined as eradication of the microorganism from the bloodstream (negative blood cultures).
Time Frame: Within 7 days from initiating the study drug
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Daptomycin 6 mg/kg IV
Number analyzed (Participants) | 37
Participants | 34

5. Secondary Outcome: Relapse
Description: Number of participants with relapse was defined as the recurrence of bacteremia within the first 3 months.
Time Frame: Within 3 months from initiating the study drug
Population: Of the 38 participants analyzed, one participant was excluded from the analyses because of microbiological failure.
Measure: Count of Participants; unit: Participants
Arm/Group | Daptomycin 6 mg/kg IV
Number analyzed (Participants) | 37
Participants | 3

6. Secondary Outcome: Number of Participants With Overall Response
Description: Overall response = symptom resolution within 3 days (since using antibiotic) + microbiological resolution within 3 days + no infection-related death + no infection-related late complications + no relapse. Infection-related late complication was defined as the development of deep-seated infection that was not present or suspected at the onset of bacteremia but was subsequently diagnosed after 1 week from initiation of study drug.
Time Frame: Within 3 days from initiating the study drug
Population: Of the 38 participants analyzed, one participant was excluded from the analyses because the date of symptom resolution was unknown.
Measure: Count of Participants; unit: Participants
Arm/Group | Daptomycin 6 mg/kg IV
Number analyzed (Participants) | 37
Participants | 25

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) and Serious Adverse Events (SAEs) were evaluated from the time of the first infusion of study drug through the end of the post-treatment visit, up to 2 years
Arm/Group | Daptomycin 6 mg/kg IV
All-Cause Mortality (participants affected / at risk) | 4/38
Serious Adverse Events (participants affected / at risk) | 18/38
Other Adverse Events (participants affected / at risk) | 18/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Daptomycin 6 mg/kg IV (N=38)
Increased Creatinine kinase (Metabolism and nutrition disorders) | 18
Rash (Skin and subcutaneous tissue disorders) | 18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Daptomycin 6 mg/kg IV (N=38)
Confusion (Nervous system disorders) | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes